CLINICAL TRIAL: NCT06584292
Title: Comparison of Caudal Block and Retrolaminar Block for Postoperative Analgesia in Concurrent Circumcision and Low Abdominal Surgery in Pediatric Patients: A Double-blind, Randomized Controlled Trial
Brief Title: Comparison of Caudal Block and Retrolaminar Block for Circumcision
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: we couldn't find enough patient.
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Engin Ihsan Turan, principal investigator, Kanuni Sultan Suleyman Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: retrolaminar blok
Record Dates: First submitted 2024-09-02; First posted 2024-09-04 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Regional Anesthesia
Keywords: Caudal block; Retrolaminar block; postoperative pain management

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The nurse was blinded to the face, legs, activity, cry, and consolability (FLACC) scores. An anesthesiologist was blinded to data collection regarding analgesic requirement and postoperative complications. Transparent sterile drapes were applied to the injection sites, and both blocks were administered to all patients to evaluate postoperative complications. Thus, the anesthetist was blinded to the postoperative complications.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Caudal block (Active Comparator): Caudal Block (CB) will applied to the patients.
  Interventions: Procedure: caudal block
- Retrolaminar Block (Active Comparator): Retrolaminar Block (RL) will applied to the patients.
  Interventions: Procedure: Retrolaminar block

INTERVENTIONS:
Procedure: caudal block — Caudal Block (CB) Procedure: The sacral hiatus was identified using an out-of-plane transverse ultrasound view at the level of the sacral cornua. The probe was then rotated longitudinally to visualize the sacrococcygeal ligament and sacral bone. A block needle was inserted through the sacrococcygeal membrane into the sacral canal using the in-plane technique, and 0.125% bupivacaine was administered at a dose of 1 mL/kg, with a maximum limit of 20 mL per side.
  Arms: Caudal block
Procedure: Retrolaminar block — Retrolaminar Block (RL) Procedure: The RL block was performed with the patient in a lateral decubitus position. The ultrasound probe was positioned at the L4 vertebral level in a paramedian sagittal plane. The probe was moved medially until the vertebral laminae were visualized. The needle was inserted using the in-plane technique, advancing from the cephalad to caudal direction until it contacted the L4 lamina. A dose of 0.1 mL/kg of 0.25% bupivacaine was then injected into the retrolaminar space.
  Arms: Retrolaminar Block

SUMMARY:
Primary Outcome:

Analgesic Efficiency: The primary outcome is the comparison of the analgesic efficacy of the retrolaminar block (RL) versus caudal block (CB) based on postoperative pain scores measured by the FLACC score. This outcome aims to evaluate how effectively each block controls postoperative pain.

Secondary Outcomes:

Analgesic Requirements:

The amount of analgesic required within the first 24 hours postoperatively. The time to the first analgesic requirement. These will be recorded during postoperative follow-up visits at 30 minutes, 1, 2, 4, 6, 12, and 24 hours by an anesthesiologist who is blinded to the study groups.

Postoperative Complications:

Urinary Retention: Defined as a distended palpable bladder associated with pain.

Motor Block: The presence of lower extremity motor block will be evaluated using the modified Bromage scale (0: No motor block; 1: Able to move the legs; 2: Unable to move the legs).

Ecchymosis and Hematoma: The presence of ecchymosis (discoloration of the skin due to blood infiltration in the subcutaneous tissues) and hematoma (abnormal swelling or hardening caused by the accumulation of blood) at the injection site will be assessed.

DETAILED DESCRIPTION:
This study is a double-blind, randomized controlled trial designed to compare the analgesic efficacy and safety of the retrolaminar block (RL) versus the caudal block (CB) in pediatric patients undergoing concurrent circumcision and lower abdominal surgery. The trial adheres to the ethical principles outlined in the Declaration of Helsinki and was conducted in the Anesthesiology and Reanimation department of a tertiary education and research hospital.

Study Population The study included pediatric patients aged 1 to 7 years who were classified as American Society of Anesthesiologists (ASA) physical status I or II. These patients were scheduled for elective, unilateral lower abdominal surgery (such as orchiopexy or hydrocelectomy) combined with circumcision. The inclusion criteria ensured the selection of otherwise healthy children with no significant comorbidities. Exclusion criteria included patients younger than 1 year or older than 7 years, those with neurological deficits, bleeding disorders, allergy to local anesthetics, infection at the injection site, congenital spinal anomalies, intellectual disabilities, psychiatric disorders, liver and/or kidney diseases, and those who declined to participate.

Randomization and Blinding Participants were randomly assigned to one of two groups (RL block or CB block) using a computer-generated randomization table. The randomization process was designed to ensure an equal distribution of patients across both groups. Both patients and the healthcare professionals involved in postoperative care were blinded to the type of block administered. To maintain blinding, both blocks were performed under sterile conditions, and identical transparent drapes were used to cover the injection sites. An anesthesiologist who was not involved in the block administration was responsible for data collection related to postoperative analgesic requirements and complications.

General Anesthesia Protocol All patients received 0.5 mg/kg of oral midazolam as premedication. In the operating room, standard monitoring was applied, and anesthesia was induced with intravenous (IV) propofol (2 mg/kg) and fentanyl (0.5 µg/kg). After the loss of the eyelash reflex, an appropriately sized laryngeal mask airway (LMA) was placed without the use of neuromuscular blocking agents. Anesthesia was maintained with sevoflurane (2%) in a mixture of 50% oxygen and air. Demographic data, including age, weight, type of surgery, duration of the procedure, and any complications, were recorded.

Regional Anesthesia Procedure Following the induction of general anesthesia and airway management, the patients were placed in the left lateral decubitus position for the regional block procedure. All blocks were performed by a single experienced operator skilled in pediatric ultrasound-guided regional anesthesia, using a 22-G, 50-mm echogenic needle. The ultrasound guidance was provided by a high-frequency (6.5-18 MHz) linear probe.

Caudal Block (CB) Procedure: The sacral hiatus was identified using an out-of-plane transverse ultrasound view at the level of the sacral cornua. The probe was then rotated longitudinally to visualize the sacrococcygeal ligament and sacral bone. A block needle was inserted through the sacrococcygeal membrane into the sacral canal using the in-plane technique, and 0.125% bupivacaine was administered at a dose of 1 mL/kg, with a maximum limit of 20 mL per side.

Retrolaminar Block (RL) Procedure: The RL block was performed with the patient in a lateral decubitus position. The ultrasound probe was positioned at the L4 vertebral level in a paramedian sagittal plane. The probe was moved medially until the vertebral laminae were visualized. The needle was inserted using the in-plane technique, advancing from the cephalad to caudal direction until it contacted the L4 lamina. A dose of 0.1 mL/kg of 0.25% bupivacaine was then injected into the retrolaminar space.

Both blocks were administered bilaterally, and the patients were repositioned supine 15 minutes before the start of the surgery.

Postoperative Monitoring and Follow-up Postoperative monitoring included heart rate, non-invasive blood pressure, and peripheral oxygen saturation. These parameters were recorded before and after the block every 5 minutes. The effectiveness of the block was assessed based on changes in heart rate and blood pressure following the surgical incision. An increase of 20% or more in these values was considered indicative of an unsuccessful block, in which case a rescue dose of fentanyl (0.5 µg/kg IV) was administered.

In the recovery room and at the ward, postoperative pain was evaluated using the FLACC scale at predefined intervals (30 minutes, 1, 2, 4, 6, 12, and 24 hours). The requirement for rescue analgesia was based on the FLACC scores, with IV paracetamol administered for scores of 2 to 4, and IV tramadol for scores above 4. Additionally, postoperative complications such as urinary retention, motor block, and the presence of ecchymosis or hematoma at the injection site were documented by the anesthesiologist blinded to the block type.

Data Collection and Statistical Analysis Demographic characteristics, surgical details, analgesic requirements, and postoperative complications were systematically recorded. The data were analyzed using IBM SPSS Statistics for Windows, Version 22.0. Normality of data distribution was assessed using the Shapiro-Wilk test, and appropriate statistical tests were applied based on data distribution (Student's t-test for normally distributed data, Mann-Whitney U test for non-parametric data, and Chi-square or Fisher's exact test for categorical data). Effect sizes were calculated using the Cohen method, and a p-value of less than 0.05 was considered statistically significant.

Randomization and Blinding Randomization was performed using a computer-generated randomization table (http://www. random.org), and patients were divided into two groups: RL and CB. The nurse was blinded to the face, legs, activity, cry, and consolability (FLACC) scores. An anesthesiologist was blinded to data collection regarding analgesic requirement and postoperative complications. Transparent sterile drapes were applied to the injection sites, and both blocks were administered to all patients to evaluate postoperative complications. Thus, the anesthetist was blinded to the postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients aged 1 to 7 years.
* Classified as American Society of Anesthesiologists (ASA) physical status I-II.
* Scheduled for elective, unilateral lower abdominal surgery (e.g., orchiopexy or hydrocelectomy) combined with circumcision.
* Patients whose parents or legal guardians provided written informed consent.

Exclusion Criteria:

* Patients younger than 1 year or older than 7 years.
* Presence of neurological deficits.
* Bleeding disorders.
* History of allergy to local anesthetic drugs.
* Presence of redness or infection at the injection site on physical examination.
* Any congenital spinal anomalies.
* Intellectual disabilities or psychiatric disorders.
* Liver and/or kidney disease.
* Patients or their guardians who declined to participate in the study.

Ages: 1 Year to 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2022-09-27 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Analgesic Efficiency | 1 day
  The primary outcome is the comparison of the analgesic efficacy of the retrolaminar block (RL) versus caudal block (CB) based on postoperative pain scores measured by the Face, Legs, Activity, Cry, Consolability (FLACC) scale. The FLACC scale is used to assess pain in pediatric patients, with scores ranging from 0 to 10. A score of 0 indicates no pain, while a score of 10 represents severe pain. Therefore, higher scores indicate worse pain outcomes. This outcome aims to evaluate how effectively each block controls postoperative pain.

SECONDARY OUTCOMES:
Analgesic Requirements: | 1 day
  The amount of analgesic required within the first 24 hours postoperatively. The time to the first analgesic requirement. These will be recorded during postoperative follow-up visits at 30 minutes, 1, 2, 4, 6, 12, and 24 hours by an anesthesiologist who is blinded to the study groups.
Postoperative Complications: | 1 day
  Urinary Retention: Defined as a distended palpable bladder associated with pain.
  Motor Block: The presence of lower extremity motor block will be evaluated using the modified Bromage scale (0: No motor block; 1: Able to move the legs; 2: Unable to move the legs).
  Ecchymosis and Hematoma: The presence of ecchymosis (discoloration of the skin due to blood infiltration in the subcutaneous tissues) and hematoma (abnormal swelling or hardening caused by the accumulation of blood) at the injection site will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Volkan Özen, Associate Proffesor, Study Chair — Health Science University İstanbul Prof Dr Cemil Taşcıoğlu City Hospital
Locations (1):
- Health Science University İstanbul Prof Dr Cemil Taşcıoğlu City Hospital, Istanbul, Okmeydanı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided